CLINICAL TRIAL: NCT04162119
Title: Safety and Efficiency Study of BCMA-PD1-CART Cells in Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanshun Wang, Chief of Hematology Department of Hainan Hospital of PLA General Hospital; Vice Chief of Hematology Department of PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNYY-XYK-01
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: BCMA; Myeloma; PD-1; Immunotherapy; Plasmocytoma; Chimeric antigen receptor T cell; Chimeric antigen receptor; B cell maturation antigen
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Plasmacytoma

STUDY DESIGN:
Intervention Model Description: This study was a single-center, open-label, single-arm, non-randomized clinical trial, which was divided into 3 groups by infusion dose level. Firstly, each dose group has 3 patients. The pretreatment regimen of cyclophosphamide (25mg/m2 for 3 consecutive days) and fludarabine (10mg/kg for 3 consecutive days) was given before CART cells were reinfused. CART cells were reinfused on the third day after the pretreatment. If no serious side effects emerges in the group, then the next group uses the subsequent higher dose. If serious side effects emerges in a single patient in any dose level, 3 more patients will be enrolled to the same dose level. After 9 or more patients, we select the safest dose and recruit more patients for CART test to explore its effectiveness.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multiple myeloma (Experimental): This study is to evaluate the efficacy and safety of BCMA-PD1-CART cells therapy for patients with Relapsed/Refractory Multiple Myeloma.
  Interventions: Biological: BCMA-PD1-CART Cell

INTERVENTIONS:
Biological: BCMA-PD1-CART Cell — This study was a single-center, open-label, single-arm, non-randomized clinical trial, which was divided into 3 groups by infusion dose level. Firstly, each dose group has 3 patients. The pretreatment regimen of cyclophosphamide (25mg/m2 for 3 consecutive days) and fludarabine (10mg/kg for 3 consecutive days) was given before CART cells were reinfused. CART cells were reinfused on the third day after the pretreatment. If no serious side effects emerges in the group, then the next group uses the subsequent higher dose. If serious side effects emerges in a single patient in any dose level, 3 more patients will be enrolled to the same dose level. After 9 or more patients, we select the safest dose and recruit more patients for CART test to explore its effectiveness.

SUMMARY:
This is a single center, non-randomized, open-label, phase 2 study to evaluate the efficacy and safety of BCMA-PD1-CART cells therapy for patients with relapsed/refractory Multiple Myeloma.

DETAILED DESCRIPTION:
Previous studies have found that multiple myeloma cells express PD-L1 at a high level. Therefore, the combination of anti-PD-1 or PD-L1 antibodies with CART therapy may further improve the clinical efficacy of CART cell for multiple myeloma.

The investigators screened PD-1 mutant that have high affinity bind with the PD-L1 ligand, and the affinity of the prepared mutant PD-1 Fc fusion protein to bind to PD-L1 reached clinical anti-PD-L1 antibody levels. The investigators prepared BCMA CART cells which secretes the mutant PD-1Fc fusion protein, and the prepared CART cell culture supernatant can well block the binding of PD-L1 to PD-1. Preclinical studies have shown that BCMA CART cells secreting mutant PD-1Fc fusion protein have a superior killing effect on PD-L1 positive multiple myeloma tumor cells to BCMA CART cells which does not express PD-1 fusion protein.

The trial was conducted to explore the safety and efficacy of BCMA-PD1-CART cells in Relapsed/Refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 14 to 80 years (including 14 and 80 years old).
2. The diagnosis was Refractory/relapsed multiple myeloma.(Meeting 1 of the follow 3 items)

   A.Primary treatment patients with no effect after first and second line treatment.

   B.Patients who relapsed after complete remission and failed to respond to two kind of therapy.

   C.the predicted survival is more than three months.
3. Flow cytometry or immunohistochemistry showed BCMA positive in tumor cells.
4. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.
5. No serious concomitant disease and major organ function is not serious abnormal.
6. No serious concomitant disease and major organ function is not serious abnormal.
7. the test meets the following indicators:

A.ALT/AST < 2.5 times the upper limit of normal (ULN) and total bilirubin≤34.2μmol/L.

B.WBC≥2.5×109/L.

C.PT/INR < 1.7 or PT was extended by less than 4 seconds.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Transduced positive T lymphocytes < 5% or amplified against CD3/CD28 stimulation < 5 times.
3. Active hepatitis B or hepatitis C, HIV/AIDS infection, any uncontrolled active infection.
4. Patients who are using steroid drugs throughout the body currently.
5. Patients who have received any gene therapy in the past.
6. Patients who are allergy to immunotherapy and related drugs.
7. Patients with heavy heart disease or poorly controlled high blood pressure.
8. Patients who received chemotherapy or radiation 4 weeks before the study began.
9. Patients who are participating in other clinical trials.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 3 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Overall Remission Rate(ORR) of BCMA-PD1-CART cells in Lymphoma | 3 years
  ORR will be assessed from the first CAR-T cell infusion to death or last follow-up
Overall survival(OS) of BCMA-PD1-CART cells in Lymphoma | 3 years
  OS will be assessed from the first CAR-T cell infusion to death or last follow-up
Progress-free survival(PFS) of BCMA-PD1-CART cells in Lymphoma | 3 years
  PFS will be assessed from the first CAR-T cell infusion to death or last follow-up
Rate of BCMA-PD1-CARTcells in peripheral blood cells | 3 years
  In vivo (peripheral blood) rate of BCMA-PD1-CARTcells were determined by means of flow cytometry.
Quantity of BCMA-PD1-CART cells copies in peripheral blood cells. | 3 years
  In vivo (peripheral blood) quantity of BCMA-PD1-CART cells copies copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Quanshun Wang, Study Chair — Hainan Hospital of Chinese PLA General Hospital; Wenshuai Zheng, Study Director — Hainan Hospital of Chinese PLA General Hospital; Lixun Guan, Study Director — Hainan Hospital of Chinese PLA General Hospital; Lu Wang, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Yuanyuan Xu, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Zhenyang Guan, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital
Locations (1):
- Hainan Hospital of Chinese PLA General Hospital, Sanya, Hainan, China

IPD SHARING:
Plan to Share IPD: No